CLINICAL TRIAL: NCT05402644
Title: Clinically Significant Portal Hypertension (CSPH) on Early-stage HCC Following Hepatectomy: What's the Impact?
Brief Title: Hepatectomy for Early-stage HCC Patients With CSPH
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CXPJJH11800001-2018306
Record Dates: First submitted 2022-05-26; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2021-05

CONDITIONS: HCC; Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-CSPH: BCLC stage A patients who underwent hepatectomy in the group without clinically significant portal hypertension (Non-CSPH)
  Interventions: Procedure: hepatectomy
- CSPH: BCLC stage A patients who underwent hepatectomy in the group with clinically significant portal hypertension (CSPH)
  Interventions: Procedure: hepatectomy

INTERVENTIONS:
Procedure: hepatectomy — Liver resection

SUMMARY:
Clinically significant portal hypertension (CSPH) can affect the surgical prognosis of early-stage (BCLC stage A) HCC. An additional stage, such as the BCLC stage A-B, can be considered.

ELIGIBILITY:
Inclusion Criteria:

HCC was diagnosed by two experienced pathologists in Child-Pugh grade A/B negative resection margin Initial diagnosis of HCC in the patients

Exclusion Criteria:

Distant transfer Not HCC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 311 HCC patients treated from December 2009 to January 2017.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2009-12-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
death | 2009--2025
  Patient survival time after surgery
recurrence | 2009--2025
  Patient recurrence time after surgery

IPD SHARING:
Plan to Share IPD: Undecided